CLINICAL TRIAL: NCT02823496
Title: Human Photoallergy Test
Brief Title: 18349-Human Photoallergy Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 18349
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): All subjects are patched with the same product
  Interventions: Other: Sunscreen Lotion , BAY 987521; Other: Untreated skin

INTERVENTIONS:
Other: Sunscreen Lotion , BAY 987521 — 50 μl/ cm2 of the test article is applied directly to two sites on the skin and covered with the appropriate patch. 24 hours later, the patches are removed. The test sites are lightly wiped with a dry cloth/tissue and 3μl/cm2 of test article is reapplied directly to the skin of the test site designated for irradiation, and lightly spread over the test site. 48 hours later the procedure is repeated to the same test sites. This process is repeated twice weekly for a total of six exposures. Formulation A: Y49-103, Formulation B: Y71-150.
Other: Untreated skin — One site is patched without treatment as control

SUMMARY:
To evaluate the potential of a test material to produce a photoallergic response.

ELIGIBILITY:
Inclusion Criteria:

* be male or female between the ages of 18 and 60 inclusive;
* be lightly pigmented (Fitzpatrick Skin Type I, II, III);
* have read and signed the written Informed Consent Form and have completed a Health Insurance Portability and Accountability Act (HIPAA) Authorization Form in conformance with 45CFR Parts 160 and 164;
* be in general good health as determined by the subject's medical history and in the discretion of the investigator;

Exclusion Criteria:

* have a visible sunburn;
* have a history of sun hypersensitivity/photosensitivity or photosensitive dermatoses;
* have a known hypersensitivity or allergy against any of the active and non-active ingredients of the investigational products.
* subjects who are employees of the CRO and/or Bayer or is a household member of an employee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Intensity of skin reactions is evaluated by 5 point scale | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Piscataway, New Jersey, United States